CLINICAL TRIAL: NCT00488839
Title: A Double-Blind, Randomized, Placebo- and Active Comparator- Controlled, Parallel Group, Multinational Study to Evaluate the PK and PD of IPX056 in Subjects With Established Spasticity Resulting From Multiple Sclerosis
Brief Title: IPX056 in Subjects With Established Spasticity Resulting From Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IPX056-B06-03; 2007-000236-16 (EudraCT Number)
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2017-02

CONDITIONS: Multiple Sclerosis
Keywords: Spasticity; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- IPX056 20 mg - OLE (Other): A single dose of IPX056 20 mg, Placebo IPX056 40 mg and Placebo Baclofen Tablet (Part 1), 9 week Open label extension of IPX056 (flexible dose design, IPX056 10 mg, IPX056 20 mg, IPX056 30 mg, IPX056 35 mg, or IPX056 40 mg)
  Interventions: Drug: IPX056 20 mg; Drug: IPX056 40 mg; Drug: Encapsulated Baclofen 20 mg; Drug: Placebo Baclofen Tablet; Drug: IPX056 10 mg; Drug: IPX056 30 mg; Drug: IPX056 35 mg; Drug: Placebo IPX056 40 mg
- IPX056 40 mg - OLE (Other): A single dose of IPX056 40 mg, Placebo IPX056 20 mg and Placebo Baclofen Tablet (Part 1), 9 week Open label extension of IPX056 (flexible dose design, IPX056 10 mg, IPX056 20 mg, IPX056 30 mg, IPX056 35 mg, or IPX056 40 mg)
  Interventions: Drug: IPX056 20 mg; Drug: IPX056 40 mg; Drug: Encapsulated Baclofen 20 mg; Drug: Placebo Baclofen Tablet; Drug: IPX056 10 mg; Drug: IPX056 30 mg; Drug: IPX056 35 mg; Drug: Placebo IPX056 20 mg
- Baclofen 20 mg - OLE (Other): A single dose of Encapsulated Baclofen 20 mg, Placebo IPX056 20 mg and Placebo IPX056 40 mg (Part 1), 9 week Open label extension of IPX056 (flexible dose design, IPX056 10 mg, IPX056 20 mg, IPX056 30 mg, IPX056 35 mg, or IPX056 40 mg)
  Interventions: Drug: IPX056 20 mg; Drug: IPX056 40 mg; Drug: Encapsulated Baclofen 20 mg; Drug: IPX056 10 mg; Drug: IPX056 30 mg; Drug: IPX056 35 mg; Drug: Placebo IPX056 20 mg; Drug: Placebo IPX056 40 mg
- Placebo - OLE (Other): A single dose of Placebo Baclofen Tablet, Placebo IPX056 20 mg and Placebo IPX056 40 mg (Part 1), 9 week Open label extension of IPX056 (flexible dose design,IPX056 10 mg, IPX056 20 mg, IPX056 30 mg, IPX056 35 mg, or IPX056 40 mg)
  Interventions: Drug: IPX056 20 mg; Drug: IPX056 40 mg; Drug: Encapsulated Baclofen 20 mg; Drug: Placebo Baclofen Tablet; Drug: IPX056 10 mg; Drug: IPX056 30 mg; Drug: IPX056 35 mg; Drug: Placebo IPX056 20 mg; Drug: Placebo IPX056 40 mg

INTERVENTIONS:
Drug: IPX056 20 mg — IPX056 Extended Release capsule containing 20 mg baclofen
  Other Names: Baclofen ER 20 mg
Drug: IPX056 40 mg — IPX056 Extended Release capsule containing 40 mg baclofen
  Other Names: Baclofen ER 40 mg
Drug: Encapsulated Baclofen 20 mg — Baclofen 20mg tablet was encapsulated for blinding.
  Other Names: Active comparator
Drug: Placebo Baclofen Tablet — Placebo capsule encapsulated placebo Baclofen tablet
  Arms: IPX056 20 mg - OLE; IPX056 40 mg - OLE; Placebo - OLE
Drug: IPX056 10 mg — IPX056 Extended Release capsule containing 10 mg baclofen
  Other Names: Baclofen ER 10 mg
Drug: IPX056 30 mg — IPX056 Extended Release capsule containing 30 mg baclofen
  Other Names: Baclofen ER 30 mg
Drug: IPX056 35 mg — IPX056 Extended Release capsule containing 35 mg baclofen
  Other Names: Baclofen ER 35 mg
Drug: Placebo IPX056 20 mg — Placebo capsule for IPX056 20 mg
  Arms: Baclofen 20 mg - OLE; IPX056 40 mg - OLE; Placebo - OLE
Drug: Placebo IPX056 40 mg — Placebo capsule for IPX056 40 mg
  Arms: Baclofen 20 mg - OLE; IPX056 20 mg - OLE; Placebo - OLE

SUMMARY:
The purpose of this study is to determine the effects, both good and bad, of IPX056 on subjects and their spasticity. This study will also determine the relationship between the amount of IPX056 in blood and the effects on spasticity. Lastly, this study will determine how long IPX056 affects spasticity.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate that IPX056 reduces spasticity, measured by Ashworth score, in subjects with multiple sclerosis (MS). This study will also (1) assess the correlation between pharmacokinetic (PK) and pharmacodynamic (PD) endpoints (Ashworth score), and (2) quantify the duration of pharmacodynamic effects for IPX056 as well as marketed baclofen tablet in subjects with Multiple Sclerosis (MS) after a single dose. Additionally, the efficacy parameters, including Multiple Sclerosis Impact Scale (MSIS)-29, spasm frequency and nighttime awakening score, spasticity control, morning stiffness, and Global Assessment of Efficacy and Tolerability, will be assessed during open-label extension period. The safety of IPX056 will be monitored throughout the study.

This study consists of 2 parts: Part I (Screening Visit & Visit 1) of the study is a single-dose, double-blind, randomized, placebo- and active comparator-controlled, parallel group design containing a single 12 hour PK/PD evaluation period. Part II is an optional, approximately 9-week open-label extension study and will start during Visit 1, immediately after Visit 1 PK/PD procedures are completed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years old. If female and of childbearing potential, continuing to practice and willing to continue throughout the study with appropriate contraceptives (defined as oral, injected, or implanted contraceptives, or barrier contraception). The subject must agree to take every precaution to ensure that pregnancy will not occur during the study. Female subjects of childbearing potential must have a negative urine pregnancy test immediately prior to study entry.
* Able to understand and willing to voluntarily sign an informed consent form (ICF) and an Authorization to Use and Disclose Protected Health Information form (as required by the Health Insurance Portability and Accountability Act {HIPAA} legislation, if appropriate for the region) prior to the performance of any study-specific procedures.
* Has a negative urine drug screen at screening visit.
* Has Definite multiple sclerosis by Poser or McDonald Criteria.
* Expanded Disability Status Scale (EDSS) rating between 3.0-8.0
* Has a normal ECG and a blood pressure <160/95 mmHg (systolic)/diastolic) at screening, measured in the sitting position after approximately 5 minutes of quiet rest.
* If the subject has a history of or presence of clinically significant peptic ulcers, liver disease, diabetes mellitus, hypertension or heart disease, the subject must be on a stable treatment regimen for a minimum of 3 months prior to Screening Visit
* Wiling to wash out current medication with anti-spasticity activities, including but not limited to baclofen, benzodiazepines, clonazepam, clonidine, dantrolene, diazepam, gabapentin, and tizanidine.
* Ashworth score of 2 or more for at least one of the three lower extremity muscle groups (hip adductor, knee flexor, knee extensor) in the most affected limb and a total minimum score of 6 for four muscle groups (the above three plus plantar flexor) on both limbs (maximum total score is 32) during screening visit and at pre-dose during PK/PD Visit 1.
* Able and willing to comply with the protocol, including availability for all scheduled clinic visits

Exclusion Criteria:

* If female, the subject is:

  1. pregnant; or planning to become pregnant; or
  2. breastfeeding; or
  3. a woman of child-bearing potential (defined as post menarche and biologically capable of becoming pregnant [i.e., not surgically sterile]) who is engaged in active heterosexual relations and is not using a barrier or hormonal form of birth control (i.e. oral, injected, or implanted contraceptives).
* History of allergic or severe intolerance to baclofen.
* Did not respond to previous baclofen treatment in any formulation.
* Treated with intrathecal baclofen within the previous 6 months prior to the Screening Visit.
* Has experienced an exacerbation of MS within 6 months prior to the Screening Visit.
* Symptomatic urinary tract infection (UTI) within 4 weeks prior to the Screening Visit and more than two (2) UTI incidents within the last 6 months.
* Serum creatinine level ≥ 2 x ULN (upper limit of normal reference range) at the Screening Visit or requires dialysis.
* Liver enzyme values ≥ 2 x ULN (upper limit of normal reference range) at the Screening Visit.
* Uncontrolled peptic ulcers, liver disease, diabetes mellitus, bladder sphincter hypertonia, hypertension or heart disease.
* History of seizure or epilepsy, or is currently taking an anti-convulsant for treatment or control of seizure.
* Concomitant neurologic conditions causing spasticity (e.g. stroke, cerebral palsy, traumatic brain injury) or rigidity (e.g. Parkinson's disease).
* Any medical condition, including psychiatric disease, which would interfere with the interpretation of the study results, the conduct of the study, or the safety of the subject.
* Currently taking antipsychotics, CNS depressants or CNS depression producing medications (including alcohol, sedating antihistamines, barbiturates, narcotics, and phenothiazines), monoamine oxidase inhibitors (MAOI, including furazolidone, procarbazine, selegiline, and tranylcypromine), and tricyclics.
* Unable or unwilling to wash out current anti-spasticity medications, including but not limited to baclofen, benzodiazepines, clonazepam, clonidine, dantrolene, diazepam, gabapentin, and/or tizanidine for Day 1, Visit 1, procedures. However, these medications will be allowed during open label study.
* Unable or unwilling to participate 12-hour PK/PD procedures during Visit 1.
* Treated with Botulinum Toxin Type A or B within the previous 6 months, or Phenol or therapeutic alcohol nerve block within 12 months prior to the Screening Visit.
* History of alcohol abuse or use of recreational drugs within 12 months prior to the Screening Visit.
* Has received an investigational drug or device within 30 days prior to the Screening Visit.
* Has clinically significant limitation of passive range of motion around any of the joints being assessed in this study.
* Has had major surgery within 3 months prior to Screening visit that may affect spasticity assessments such as abdominal surgery, back surgery, lower leg and knee surgeries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Overall mean changes from predose (baseline) in total Ashworth scores of the four lower extremity muscle groups (hip adductors, knee flexors, knee extensors, and plantar flexors) of both lower limbs over 12 hours assessed hourly after dosing | 12 hours

SECONDARY OUTCOMES:
Duration of effect (improvement in Ashworth Scale) for IPX056 | 12 hours
Establishment of relationships between baclofen plasma concentration with improvement in Ashworth Scale | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Impax Study Director, Study Director — Impax Laboratories, LLC
Locations (31):
- United States (20):
  - Northwest NeuroSpecialists, Tucson, Arizona
  - OrthoArkansas, P. A., Little Rock, Arkansas
  - OrthoArkansas, P.A., Little Rock, Arkansas
  - Patricia Fodor, Colorado Springs, Colorado
  - Sunrise Clinical Research, Hollywood, Florida
  - Meridien Research, Tampa, Florida
  - MS Center of Atlanta, Atlanta, Georgia
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Elkhardt Clinic, Elkhart, Indiana
  - MidAmerica Neuroscience Institute, Lenexa, Kansas
  - Springfield Neurology, Springfield, Massachusetts
  - General Clinical Research Center 7A, Ann Arbor, Michigan
  - Medex Healthcare Research, Inc., Saint Louis, Michigan
  - Northern Michigan Neurology, Traverse City, Michigan
  - Winthrop University Hospital, Mineola, New York
  - Crozer Chester Medical Center, Upland, Pennsylvania
  - Bhupesh Dihenia, Lubbock, Texas
  - Integra Clinical Research, San Antonio, Texas
  - Neurological Research Center, Bennington, Vermont
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
- Canada (2):
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - Foothills Medical Centre, MS Clinic, SSB, Calgary
- West-Tallinn Central Hospital, Tallinn, Estonia
- Vecmilgravis Hospital, Latvian Maritime Medicine Center, Riga, Latvia
- Ukraine (7):
  - Chernihiv Regional Hospital Department of Neurology, Chernihiv
  - Neurology and Neurosurgery Dpt., Postgraduation training faculty, Dnipropetrovsk State medical Academy, Dnipropetrovsk
  - Institue of Neruology, Psychiatry and Narcology of AMS of Ukraine, Kharkiv
  - Department of nervous system demyelization diseases of City Clinical Hospital, Kyiv
  - Odessa Regional Clinical Hospital, Odesa
  - Neurology department of Ukraine medical stomatological akademy, Poltava
  - Vinnytsya Regional Psychoneurological Hospital, Vinnytsia

IPD SHARING:
Plan to Share IPD: No